CLINICAL TRIAL: NCT01552408
Title: A Phase I/II, Randomized, Study for Diabetic Macular Edema Using 0.3mg Ranibizumab Combined With Targeted PRP Monthly for 4 Months,Then PRN vs. 0.3mg Ranibizumab 4 Months Monotherapy, Then as Needed(DME-AntiVEgf) DAVE
Brief Title: Efficacy & Safety Trial of Intravitreal Injections Combined With PRP for CSME Secondary to Diabetes Mellitus (DAVE)
Acronym: DAVE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David M. Brown, M.D. (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, David M. Brown, M.D., Director Greater Houston Retina Research, Greater Houston Retina Research
Organization: Greater Houston Retina Research (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML27954
Record Dates: First submitted 2012-02-28; First posted 2012-03-13 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Macular Edema
Keywords: Non Proliferative Diabetic Retinopathy; Diabetic Retinopathy; Macular Edema; Background Diabetic Retinopathy; Pre Proliferative Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy; Macular Edema | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.3 mg Ranibizumab (Active Comparator): Cohort 1: Subjects will receive 4 IVT of 0.3 mg ranibizumab every 28 days (+/- 7 days), then will be seen monthly (+/- 7 days) & will receive IVT of 0.3 mg ranibizumab on a pro re nata (PRN) schedule per retreatment criteria.
  Interventions: Drug: 0.3 mg ranibizumab
- Targeted PRP with 0.3 mg Ranibizumab (Experimental): Cohort 2: Subjects will receive 4 it of 0.3 mg ranibizumab every 28 days (+/- 7 days), then will then be seen monthly (+/- 7 days) & receive IVT of 0.3 mg ranibizumab on a PRN schedule per retreatment criteria based on the evaluating Investigator's assessment of disease activity. In addition, at Day 7 they will receive targeted pan-retinal photocoagulation (PRP) based on ultra wide field angiography. Ultra wide field angiography will be performed every 3 months to indicate areas of peripheral ischemia, which will be selectively be treated with PRP at Month 6, Month 18, and Month 25, preserving areas of more perfused retina.
  Interventions: Drug: 0.3 mg ranibizumab; Procedure: Targeted Pan Retinal Photocoagulation

INTERVENTIONS:
Drug: 0.3 mg ranibizumab — Cohort 1: Subjects will receive 4 mandatory intravitreal injections of 0.3 mg ranibizumab every 28 days (+/- 7 days). They will then be seen monthly (+/- 7 days) and will receive intravitreal injections of 0.3 mg ranibizumab on a PRN schedule per retreatment criteria based on the evaluating Investigator's assessment of disease activity.
  Other Names: Lucentis
Procedure: Targeted Pan Retinal Photocoagulation — Cohort 2: Subjects will receive 4 mandatory intravitreal injections of 0.3 mg ranibizumab every 28 days (+/- 7 days). They will then be seen monthly (+/- 7 days) and will receive intravitreal injections of 0.3 mg ranibizumab on a PRN schedule per retreatment criteria based on the evaluating Investigator's assessment of disease activity. In addition, at V3 (Day 7) they will receive targeted pan retinal photocoagulation (PRP) based on ultra wide 200º field angiography. After the first session of PRP, subject's will have ultra wide 200º field angiography performed every 3 months to indicate areas of peripheral ischemia, which will be selectively treated at V9 (Month 6), V21 (Month 18), and V28 (Month 25), preserving areas of more perfused retina. This will minimize any visual field loss secondary to nonselective pan-retinal photocoagulation.
  Other Names: PRP; Laser Photocoagulation; Pan Retinal Photocoagulation
  Arms: Targeted PRP with 0.3 mg Ranibizumab

SUMMARY:
This study is a Phase I/II, multicenter, randomized, study of the efficacy and safety of ranibizumab injection monotherapy verses a duel therapy of 0.3mg ranibizumab combined with ultra wide, 200° field angiography guided pan retinal photocoagulation in patients with CSME-CI secondary to diabetes mellitus (Type 1 or 2).

DETAILED DESCRIPTION:
Approximately 40 eyes will be randomized at 3 investigational centers in the United States. This study consists of a screening period of up to 14 days (Days -14 to -1), and a 36-month treatment period (Day 0 to Month 36). Subjects who provide consent will enter the screening period to determine eligibility. As part of the screening process, the examining investigator will evaluate the macular foveal avascular zone fluorescein images to determine subjects' eligibility. Eligible subjects will be randomized in a 1:1 ratio so that approximately 20 eyes will receive 0.3 mg ranibizumab monotherapy, and approximately 20 eyes will receive 0.3 mg ranibizumab combined with Ultra wide 200° field angiogram guided targeted pan retinal photocoagulation (PRP). Subjects must meet VA and retinal thickness eligibility requirements during the screening period. The subject can have both eyes in the study. If both eyes are eligible, one eye will be randomized, to cohort 1 while the other eye will be randomized to the cohort 2. A subject with both eyes in the trial will have each eye in a separate cohort.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide signed informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization.
* Age ≥ 18 years
* Diabetes Mellitus (Type 1 or 2). The following will be considered as sufficient evidence that diabetes is present:

  * Current regular use of insulin for the treatment of diabetes
  * Current regular use of oral antihyperglycemic agents for the treatment of diabetes
  * Documented diabetes according to the American Diabetes Association and/or World Health Organization criteria.
* BCVA score in the study eye of 20/32 to 20/320 approximate snellen equivalent using the ETDRS protocol at an initial testing distance of 4 meters, confirmed by the investigator.
* High Definition OCT (Spectralis) central retinal thickness measurement of ≥ 300 µm
* Decrease in visual acuity is determined to be primarily the result of DME and not to other cause.
* Ability and willingness to return for all scheduled visits and assessments.
* Clear ocular media and adequate pupillary dilatation to permit good quality fundus photography.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from this study:

General Exclusion Criteria

* Pregnancy (positive pregnancy test) or lactation
* Sexually active women of childbearing potential* who are unwilling to practice adequate contraception or abstinence during the study. (*Although no birth control method is 100% effective, the following are considered adequate means of contraception: surgical sterilization, use of oral contraceptives, barrier contraception using either a condom or diaphragm with spermicidal gel, intrauterine devices, or contraceptive hormone implants or patches. A subject's primary care physician, obstetrician, or gynecologist should be consulted regarding an appropriate form of birth control)
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial] Ocular Exclusion Criteria
* Prior Ocular Treatment:

  * History of vitrectomy surgery in the study eye
  * Any pan-retinal photocoagulation in the study eye
  * Prior treatment with intraocular or subconjunctival steroids in the study eye 4 months prior to screen
  * Previous treatment with antiangiogenic drugs in either eye (pegaptanib sodium, anecortave acetate, bevacizumab, ranibizumab, etc.) within 2 months of Day 0 visit
  * Systemic corticosteroids 4 months prior to screen

Concurrent Ocular Conditions:

* Any concurrent ocular condition in the study eye (e.g., cataract or age-related macular degeneration) that, in the opinion of the investigator could: require medical or surgical intervention during the study period to prevent or treat visual loss that might result from that condition; or, if allowed to progress untreated, could likely contribute to a loss of at least 2 Snellen equivalent lines of BCVA over the study period
* Active intraocular inflammation (grade trace or above) in the study eye
* Current vitreous hemorrhage in the study eye
* History of rhegmatogenous retinal detachment or macular hole (Stage 3 or 4) in the study eye
* Active infectious conjunctivitis, keratitis, scleritis, or endophthalmitis in either eye
* Aphakia or absence of the posterior capsule in the study eye
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Day 0
* Uncontrolled glaucoma in the study eye (defined as IOP ≥ 30 mmHg despite treatment with anti-glaucoma medication)
* History of glaucoma-filtering surgery in the study eye
* History of corneal transplant in the study eye
* High Risk PDR: New vessels within one disc diameter of the optic nerve head that are larger than one-third disc area
* Vitreous or preretinal hemorrhage associated with less extensive NVD or with NVE one-half disc area or more in size
* Extensive damage to the fovea vascular zone as determined by the principal investigator or designated site personnel
* Spherical equivalent of the refractive error in the study eye of more that -8.00 diopter of myopia
* Vitreomacular traction (vitreomacular attachment ok) Concurrent Systemic Conditions
* Uncontrolled blood pressure (defined as systolic > 180 mmHg and/or diastolic > 110 mmHg while patient is seated. *If a subject's initial reading exceeds these values, a second reading may be taken 30 or more minutes later. If the subject's blood pressure needs to be controlled by antihypertensive medication, the subject can become eligible if medication is taken continuously for at least 30 days prior to Day 0
* Atrial fibrillation not managed by subject's primary care physician or cardiologist within 3 months of screening visit
* History of stroke within the last 3 months of screening visit
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or renders the patient at high risk for treatment complications
* Current treatment for active systemic infection
* Active malignancy
* History of allergy to fluorescein, not amenable to treatment
* Inability to obtain fundus photographs or fluorescein angiograms of sufficient quality to be analyzed and graded.
* Previous participation in any studies of investigational drugs within 1 month preceding Day 0 (excluding vitamins and minerals)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-05-18 (Actual); Study Completion 2017-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Brown, MD, Principal Investigator — Director Greater Houston Research
Locations (3):
- United States (3):
  - Retina Consultants of Houston, Houston, Texas
  - Retina Consultants of Houston, Katy, Texas
  - Retina Consultants of Houston, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klein R, Meuer SM, Moss SE, Klein BE. Retinal microaneurysm counts and 10-year progression of diabetic retinopathy. Arch Ophthalmol. 1995 Nov;113(11):1386-91. doi: 10.1001/archopht.1995.01100110046024. PMID 7487599
- [Background] Klein M. Prevention and treatment of the complications of diabetes mellitus. N Engl J Med. 1995 Sep 21;333(12):802. doi: 10.1056/NEJM199509213331215. No abstract available. PMID 7643896
- [Background] Cruickshanks KJ, Moss SE, Klein R, Klein BE. Physical activity and the risk of progression of retinopathy or the development of proliferative retinopathy. Ophthalmology. 1995 Aug;102(8):1177-82. doi: 10.1016/s0161-6420(95)30893-7. PMID 9097744
- [Background] Diabetic Retinopathy Clinical Research Network; Scott IU, Edwards AR, Beck RW, Bressler NM, Chan CK, Elman MJ, Friedman SM, Greven CM, Maturi RK, Pieramici DJ, Shami M, Singerman LJ, Stockdale CR. A phase II randomized clinical trial of intravitreal bevacizumab for diabetic macular edema. Ophthalmology. 2007 Oct;114(10):1860-7. doi: 10.1016/j.ophtha.2007.05.062. Epub 2007 Aug 15. PMID 17698196
- [Background] Writing Committee for the Diabetic Retinopathy Clinical Research Network; Fong DS, Strauber SF, Aiello LP, Beck RW, Callanan DG, Danis RP, Davis MD, Feman SS, Ferris F, Friedman SM, Garcia CA, Glassman AR, Han DP, Le D, Kollman C, Lauer AK, Recchia FM, Solomon SD. Comparison of the modified Early Treatment Diabetic Retinopathy Study and mild macular grid laser photocoagulation strategies for diabetic macular edema. Arch Ophthalmol. 2007 Apr;125(4):469-80. doi: 10.1001/archopht.125.4.469. PMID 17420366
- [Background] From the NIH: Study identifies four factors in diabetic retinopathy associated with high risk of severe visual loss. JAMA. 1979 Apr 13;241(15):1581. No abstract available. PMID 581885
- [Background] Four risk factors for severe visual loss in diabetic retinopathy. The third report from the Diabetic Retinopathy Study. The Diabetic Retinopathy Study Research Group. Arch Ophthalmol. 1979 Apr;97(4):654-5. doi: 10.1001/archopht.1979.01020010310003. PMID 426679
- [Background] Photocoagulation for diabetic macular edema. Early Treatment Diabetic Retinopathy Study report number 1. Early Treatment Diabetic Retinopathy Study research group. Arch Ophthalmol. 1985 Dec;103(12):1796-806. PMID 2866759
- [Background] Treatment techniques and clinical guidelines for photocoagulation of diabetic macular edema. Early Treatment Diabetic Retinopathy Study Report Number 2. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1987 Jul;94(7):761-74. doi: 10.1016/s0161-6420(87)33527-4. PMID 3658348
- [Background] Muggeo M. DCCT and us: how far are we from implementation? Acta Diabetol. 1993;30(3):115-7. doi: 10.1007/BF00572852. No abstract available. PMID 8111068
- [Background] Luddeke HJ. [Continuing education provided by the Diabetes Society. Results of the UKPDS (United Kingdom Diabetes Society) and therapeutic guidelines concerning diabetes type II]. Fortschr Med. 1998 Nov 30;116(33):35-8. No abstract available. German. PMID 9889462
- [Background] Watkins P. The UKPDS. A model for gathering the evidence for the management of chronic diseases. UK Prospective Diabetes Study Group. J R Coll Physicians Lond. 1998 Nov-Dec;32(6):510-1. No abstract available. PMID 9881303
- [Background] Diabetic Retinopathy Clinical Research Network (DRCR.net); Beck RW, Edwards AR, Aiello LP, Bressler NM, Ferris F, Glassman AR, Hartnett E, Ip MS, Kim JE, Kollman C. Three-year follow-up of a randomized trial comparing focal/grid photocoagulation and intravitreal triamcinolone for diabetic macular edema. Arch Ophthalmol. 2009 Mar;127(3):245-51. doi: 10.1001/archophthalmol.2008.610. PMID 19273785
- [Background] Scott IU, Danis RP, Bressler SB, Bressler NM, Browning DJ, Qin H; Diabetic Retinopathy Clinical Research Network. Effect of focal/grid photocoagulation on visual acuity and retinal thickening in eyes with non-center-involved diabetic macular edema. Retina. 2009 May;29(5):613-7. doi: 10.1097/IAE.0b013e3181a2c07a. PMID 19373126
- [Background] Jonas JB, Strueven V, Kamppeter BA, Harder B, Spandau UH, Schlichtenbrede F. Visual acuity change after intravitreal triamcinolone in various types of exudative age-related macular degeneration. J Ocul Pharmacol Ther. 2006 Oct;22(5):370-6. doi: 10.1089/jop.2006.22.370. PMID 17076632
- [Background] Martidis A, Duker JS, Greenberg PB, Rogers AH, Puliafito CA, Reichel E, Baumal C. Intravitreal triamcinolone for refractory diabetic macular edema. Ophthalmology. 2002 May;109(5):920-7. doi: 10.1016/s0161-6420(02)00975-2. PMID 11986098
- [Background] Audren F, Tod M, Massin P, Benosman R, Haouchine B, Erginay A, Caulin C, Gaudric A, Bergmann JF. Pharmacokinetic-pharmacodynamic modeling of the effect of triamcinolone acetonide on central macular thickness in patients with diabetic macular edema. Invest Ophthalmol Vis Sci. 2004 Oct;45(10):3435-41. doi: 10.1167/iovs.03-1110. PMID 15452046
- [Background] Aiello LP, Edwards AR, Beck RW, Bressler NM, Davis MD, Ferris F, Glassman AR, Ip MS, Miller KM; Diabetic Retinopathy Clinical Research Network. Factors associated with improvement and worsening of visual acuity 2 years after focal/grid photocoagulation for diabetic macular edema. Ophthalmology. 2010 May;117(5):946-53. doi: 10.1016/j.ophtha.2009.10.002. Epub 2010 Feb 1. PMID 20122739

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 29 unique participants were enrolled in the study. 11 of these 29 had both eyes assigned to each intervention. Therefore, a total of 40 eyes were randomized in the trial.
Units Other Than Participants: Eyes
Groups:
- 0.3 mg Ranibizumab: Subjects will receive 4 mandatory intravitreal injections of 0.3 mg ranibizumab every 28 days (+/- 7 days). They will then be seen monthly (+/- 7 days) and will receive intravitreal injections of 0.3 mg ranibizumab on a PRN schedule per retreatment criteria based on the evaluating Investigator's assessment of disease activity.
- Targeted Pan-retinal Photocoagulation With 0.3 mg Ranibizumab: Subjects will receive 4 mandatory intravitreal injections of 0.3 mg ranibizumab every 28 days (+/- 7 days). They will then be seen monthly (+/- 7 days) and will receive intravitreal injections of 0.3 mg ranibizumab on a pro re nata (PRN) schedule per retreatment criteria based on the evaluating Investigator's assessment of disease activity. In addition, at V3 (Day 7) they will receive targeted pan-retinal photocoagulation (PRP) based on ultra wide 200º field angiography (see Appendix C). After the first session of PRP, subject's will have ultra wide 200º field angiography performed every 3 months to indicate areas of peripheral ischemia, which will be selectively treated at V9 (Month 6), V21 (Month 18), and V28 (Month 25), preserving areas of more perfused retina. This will minimize any visual field loss secondary to nonselective pan-retinal photocoagulation.
Period: Overall Study
Arm/Group | 0.3 mg Ranibizumab | Targeted Pan-retinal Photocoagulation With 0.3 mg Ranibizumab
Started | 20; 20 Eyes | 20; 20 Eyes
Completed | 16; 16 Eyes | 18; 18 Eyes
Not Completed | 4; 4 Eyes | 2; 2 Eyes
Not completed — Lost to Follow-up | 2 | 0
Not completed — Relocation | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Targeted PRP With 0.3 mg Ranibizumab: Subjects will receive 4 mandatory intravitreal injections of 0.3 mg ranibizumab every 28 days (+/- 7 days). They will then be seen monthly (+/- 7 days) and will receive intravitreal injections of 0.3 mg ranibizumab on a PRN schedule per retreatment criteria based on the evaluating Investigator's assessment of disease activity. In addition, at V3 (Day 7) they will receive targeted pan-retinal photocoagulation (PRP) based on ultra wide 200º field angiography (see Appendix C). After the first session of PRP, subject's will have ultra wide 200º field angiography performed every 3 months to indicate areas of peripheral ischemia, which will be selectively treated at V9 (Month 6), V21 (Month 18), and V28 (Month 25), preserving areas of more perfused retina. This will minimize any visual field loss secondary to nonselective pan-retinal photocoagulation.
- Total: Total of all reporting groups
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab | Total
Number analyzed (Participants) | 20 | 20 | 29
Number analyzed (Eyes) | 20 | 20 | 40
Age, Customized [Mean (Full Range); unit: years]
  Age | 55 [45 to 69] | 56 [31 to 75] | 55 [31 to 75]
Sex/Gender, Customized [Number; unit: Eyes]
  Gender : Female | 4 | 5 | 9
  Gender : Male | 16 | 15 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Number of Right Eyes Enrolled [Number; unit: Eyes] | 7 | 11 | 18
Glycated Hemoglobin [Mean (Full Range); unit: Percentage] | 8.8 [5.9 to 12.9] | 8.0 [5.9 to 12.8] | 8.4 [5.9 to 12.9]
Diabetes Mellitus Diagnosis Year [Median (Full Range); unit: year] | 2002 [1982 to 2012] | 2001 [1980 to 2012] | 2001 [1980 to 2012]
Diabetic Macular Edema Diagnosis Year [Mean (Full Range); unit: year] | 2012 [2008 to 2014] | 2012 [2010 to 2014] | 2012 [2008 to 2014]
Early Treatment Diabetic Retinopathy Study Best-Corrected Visual Acuity [Mean (Full Range); unit: letters] | 59.1 [23 to 75] | 60.1 [37 to 76] | 59.6 [23 to 76]
Central Retinal Thickness [Mean (Full Range); unit: microns] | 571 [262 to 1034] | 488 [273 to 946] | 530 [262 to 1034]

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Ranibizumab Injections in Each of the Two Cohorts in a 36 Month Period
Description: Assess the number of ranibizumab injections in the ranibizumab and targeted panretinal photocoagulation (PRP) with ranibizumab cohorts through Month 36.
Time Frame: 36 Months
Population: All participants were included in analysis. Among participants who failed to complete the study, the last observation was carried forward for analysis at Month 36.
Measure: Mean (Full Range); unit: injections
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 20 | 20
injections | 24.4 [10 to 34] | 27.1 [12 to 36]

2. Primary Outcome: Mean Change Over Time in Early Treatment Diabetic Retinopathy Study Best Corrected Visual Acuity (ETDRS BCVA) Through Month 36
Description: Evaluate the mean change over time in ETDRS BCVA in the ranibizumab and targeted PRP with ranibizumab cohorts through Month 36.
Time Frame: 36 Months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 20 | 20
letters | 13.9 (10.2) | 8.2 (16.1)

3. Primary Outcome: Incidence and Severity of Ocular and Non-ocular Adverse Events (AE's) Through Month 36.
Description: Incidence and severity of ocular and non-ocular adverse events (AE's) in the monotherapy and combination cohorts through Month 36.
Time Frame: 36 Months
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 20 | 20
Participants
  Participants Experiencing Serious Ocular AE | 2 | 1
  Participants Experiencing Serious Systemic AE | 7 | 9

4. Secondary Outcome: Patients Who Experience a Loss of 15 or More Letters From Baseline to Month 12, 24, and 36 in ETDRS BCVA.
Description: Percentage of patients in the ranibizumab and targeted PRP with ranibizumab cohorts who experience a loss of 15 or more letters from Baseline to Month 12, 24, and 36 in ETDRS BCVA.
Time Frame: Month 12, 24, and 36
Population: All participants were included in analysis. Due to participant attrition and missed visits, the population analyzed at each time point is equal to or smaller than the population still enrolled at that time point.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 20 | 20
Participants
  12 Months | 0 | 0
  24 Months | 0 | 1
  36 Months | 0 | 1

5. Secondary Outcome: Determine Percentage of Patients Who Experience a Gain of 15 or More Letters From Baseline to Month 12, 24, and 36 in ETDRS BCVA
Description: Determine percentage of patients who experience a gain of 15 or more letters from Baseline to Month 12, 24, and 36 in ETDRS BCVA in the ranibizumab and targeted PRP with ranibizumab cohorts.
Time Frame: Month 12, 24, and 36
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 20 | 20
Participants
  Month 12 | 10 | 5
  Month 24 | 10 | 6
  Month 36 | 9 | 5

6. Secondary Outcome: Evaluate Mean Change in Central Retinal Thickness Over Time Through Month 12, 24, and 36 as Assessed by High Resolution OCT's.
Description: Evaluate mean change in central retinal thickness in the ranibizumab and targeted PRP with ranibizumab cohorts over time through Month 12, 24, and 36 as assessed by high resolution OCT's.
Time Frame: Month 12, 24, and 36
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 20 | 20
microns
  Month 12 | -301 (255) | -161 (188)
  Month 24 | -296 (238) | -169 (172)
  Month 36 | -302 (246) | -152 (149)

7. Secondary Outcome: Patients With Persistent Macular Edema Post-intravitreal Injection.
Description: Percentage of patients with persistent macular edema post-intravitreal injection in the ranibizumab and targeted PRP with ranibizumab cohorts.
Time Frame: Month 36
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | 0.3 mg Ranibizumab | Targeted Pan-retinal Photocoagulation With 0.3 mg Ranibizumab
Number analyzed (Participants) | 17 | 18
Participants | 9 | 12

8. Secondary Outcome: Mean Change in Peripheral Visual Field as Measured by Goldmann Visual Field at Screen and Month and 36.
Description: Mean change in peripheral visual field as measured by Goldmann visual field at screen and Month 36 in the ranibizumab and targeted PRP with ranibizumab cohorts.
Time Frame: 36 Months
Population: Participants that had poor fix (resulting in inaccurate results), missing baseline results, or missing Month 36 results were excluded.
Measure: Mean (Standard Deviation); unit: degrees squared
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
Number analyzed (Participants) | 9 | 8
degrees squared | -215 (1957) | -1723 (3532)

ADVERSE EVENTS:
Time Frame: 3 years (entire study period)
Description: Adverse events were assessed at every study visit during the 3-year trial
Arm/Group | 0.3 mg Ranibizumab | Targeted PRP With 0.3 mg Ranibizumab
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 9/20 | 10/20
Other Adverse Events (participants affected / at risk) | 12/20 | 13/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg Ranibizumab (N=20) | Targeted PRP With 0.3 mg Ranibizumab (N=20)
Neovascular glaucoma (Eye disorders) | 2 (2) | 0 (0)
Vitreous hemorrhage with acute vision loss (Eye disorders) | 0 (0) | 1 (1)
Sepsis (Immune system disorders) | 1 (1) | 1 (1)
Systolic heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Osteomyelitits (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Worsening renal failure (Renal and urinary disorders) | 3 (3) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg Ranibizumab (N=20) | Targeted PRP With 0.3 mg Ranibizumab (N=20)
Vitreous hemorrhage (Eye disorders) | 2 (2) | 2 (2)
Neovascularization elsewhere (Eye disorders) | 4 (4) | 0 (0)
Neovascularization of the disc (Eye disorders) | 2 (2) | 0 (0)
Neovascularization of the iris (Eye disorders) | 1 (2) | 0 (0)
Worsening glaucoma (Eye disorders) | 3 (3) | 0 (0)
Worsening cataract (Eye disorders) | 3 (3) | 6 (6)
Posterior vitreous detachment (Eye disorders) | 4 (4) | 5 (5)
Epiretinal membrane (Eye disorders) | 1 (1) | 3 (3)
Hyphema (Eye disorders) | 2 (2) | 0 (0)
Dilated pupil (Eye disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The key limitation is the small population size analyzed through 3 years; subject attrition due to elderly population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT01552408/Prot_SAP_000.pdf